CLINICAL TRIAL: NCT06475079
Title: Correlation Between BMI and Craniovertebral Angle and Their Impact on Hand Grip Strength and Neck Functional Disability in Egyptian University Student
Status: Not yet recruiting | Type: Observational
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Ababa, lecturer of internal physical therapy , Ahram Cadian University, Ahram Canadian University
Other Study IDs: P.T - ORT- 4/2024-540
Record Dates: First submitted 2024-06-12; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group (A):: Body mass index < 25
  Interventions: Other: • FHP app (Pyeongtaek, South Korea) mobile application
- Group (B):: Body mass index > 25
  Interventions: Other: • FHP app (Pyeongtaek, South Korea) mobile application

INTERVENTIONS:
Other: • FHP app (Pyeongtaek, South Korea) mobile application — FHP app (Pyeongtaek, South Korea) mobile application ,is mobile application to asses cranio vertebral angle
  Other Names: • Hand dynamometer; • Visual Analogue Scale; • Arabic Neck Disability Index

SUMMARY:
Objective: To find the relation between cranio-vertebral angle and hand grip strength in university student mobile users.

Design: cross sectional study. Setting: Ahram Candian University Subjects:100 male and female university students with age ranged from 20 to 30 years old will participate in this study.

Intervention: cross sectional study to detect the relation between cranio-vertebral angle and hand grip strength in university student mobile users.

Main measures:

* FHP app (Pyeongtaek, South Korea) mobile application
* Hand dynamometer (the JAMAR® Hydraulic Hand) (Lupton-Smith et al.,2022)
* Mechanical height and weight scale
* Visual Analogue Scale
* Arabic Neck Disability Index Results: The results will be obtained via one-way analyses of variance (ANOVA).

ELIGIBILITY:
Inclusion Criteria:

* • Their ages will range from 20-30 years old.

  * Their BMI will be between than 20- 30kg/m2.
  * All of them suffer from mild degree of neck pain.
  * The subjects complain from neck pain for 1 month ago
* Exclusion criteria:

Exclusion criteria were a history of any of the following condition:

* inflammatory diseases or any rheumatic disorders,
* a history of vertebral fractures
* surgical spinal fixation.
* •any neurological disorders like MS

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 100 male and female patients Their ages will range from 20-30 years old. Their BMI will be between than 20- 30kg/m2, All of them suffer from mild degree of neck pain and They complain from neck pain for 1 month ago
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-26 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
craniovertebral angle will measured by FHP (Forward Head Posture ) mobile application | baseline
  It is a mobile application which is objective to detect the cervical posture by measuring the CV angle. It is an application that requires an Android version 4.0 or higher installed on a smartphone
Hand grip strength will measured by Hand dynamometer (the JAMAR® Hydraulic Hand) | baseline
  it is tool used to asses hand grip strength
Pain level will measured by Visual Analogue Scale | base line
  VAS is a line with a length of 10 where one end (right) means no pain and the other means severe unbearable pain. Each patient was asked to put a mark on the line that mostly describe his or her pain intensity.
Neck functional disability will assess by Arabic Neck Disability Index | baseline
  it consist of 10 questions in total, including ones about pain intensity, personal care, lifting, reading, headaches, driving, concentration, work, sleeping, and recreation Each item is scored from 0 (no disability) to 5 (total disability)